CLINICAL TRIAL: NCT00866151
Title: A to Z Study Follow-up: Collection of DNA Data From Buccal Swabs
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Interleukin Genetics, Inc. (Industry)
Responsible Party: Karen Shaver / Director of Clinical Operations, Interleukin Genetics Inc.,
Other Study IDs: ILI-08-108WMGTP; 14895
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Weight Management; Diet Conditions; Dietary Recommendations; Overweight Management; Obesity
Keywords: genetic biomarker; biomarker; molecular diagnostics; genes; genetics; overweight management; weight management; weight reduction; SNPs; single nucleotide polymorphisms
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal swabs are collected by Stanford and sent to Interleukin Genetics for genotyping.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Previously enrolled subjects in the "Benefits and Risks of Alternative Weight Loss Strategies - a Clinical Trial", which was run at Stanford 2003-2005. (A to Z Study)

SUMMARY:
The goal of this study is to determine the association between genotypes and diet. The weight and weight loss data are already available from the previously completed study called: A to Z Study - Benefits and Risks of Alternative Weight Loss Strategies - A Clinical Trial, which was performed from 2003-2005 at Stanford University. In the present study, Interleukin Genetics will obtain DNA samples from the previously enrolled study subjects to investigate genetic influence of the response to macronutrient compositions of low caloric diets to weight loss.

DETAILED DESCRIPTION:
Interleukin Genetics has derived, through an extensive search of the scientific literature, a genetic test panel in the area of Weight Management (WM), which includes the genes that have been shown to affect body weight. These genes have been associated with elevated risk for obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI (body mass index): 27-40 kg/m2
* Gender: Women only
* Age: 25-50
* Menopausal status: pre-menopausal
* Weight stable for last 2-months
* Not on a weight loss plan
* No ethnic restrictions
* No plans to move from the area over the next 6-months
* Willing to accept random assignment
* Possess English speaking and reading skills to understand and complete forms such as informed consent and study evaluation

Exclusion Criteria:

* Hypertension
* Diabetes (type 1 or 2) or history of gestational diabetes
* Heart disease diagnosis
* Renal or lever disease
* Active neoplasms
* Pregnant, lactating, within 6-months of birth, or planning to become pregnant in the next 6-months
* Hyperthyroidism, unless treated and under control
* Medications known to affect weight / energy expenditure
* Excessive alcohol intake (self-reported, > 3 drinks/day)
* Postmenopausal, including surgical menopause
* Currently under psychiatric care, or severely clinically depressed (>17 on Beck Inventory)

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population for the A to Z study are premenopausal women who are overweight (BMI 27-40 kg/m2) but in otherwise good general health. Overweight participants with potentially confounding health conditions are excluded (eg., hypertension, diabetes, heart disease, cancer). Children were not included in this study. The participants were asked to agree to a random assignment to dietary plans.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-06 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
The PRIMARY objective of this study is to identify genotype-diet interaction on weight, body fat, and BMI. | 1 year

SECONDARY OUTCOMES:
The SECONDARY objective is to explore the association of single nucleotide polymorphisms (SNPs) with other metabolic parameters, such as blood lipid profile, insulin level, and other cardiovascular risk factors. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Gardner, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States